CLINICAL TRIAL: NCT02808520
Title: Social Inequalities in the Participation and Activity in Children and Adolescents With Hodgkin-lymphoma. A Prospective Multicenter Cohort Study of Social and Personal Influencing Factors
Brief Title: Social Inequalities in the Participation and Activity in Children and Adolescents With Hodgkin-lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: German Cancer Aid (Other); University of Giessen (Other)
Responsible Party: Principal Investigator, Julia Roick, MSc, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: 111412
Record Dates: First submitted 2016-06-16; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Social participation; Children and adolescents with cancer; Quality of life with hodgkin-lymphoma; Social inequalities and cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hodgkin-lymphoma: Children and adolescents aged 10-18 years

SUMMARY:
Purpose of this study is to determine the influence of social factors on participation and activity among children and adolescents aged 10-18 years with hodgkin-lymphoma. Furthermore personal and treatment-related factors and their impact on participation will be explored.

DETAILED DESCRIPTION:
Hodgkin-lymphoma is a rare malignancy among children and adolescents (about 140 each year in Germany) which is highly curable. Beside this therapeutic success, a lot of therapy-related long-term problems arise (e.g. fertility disorders, thyroid diseases, secondary malignancies). While most of the studies focused on mental and physical impairments, little attention has been drawn to social dimensions of health. Due to the disease and the requirements of the therapy, participation of children with hodgkin-lymphoma can be impaired acutely or chronically. This can be of serious consequences, because participation in daily life is an important component of the development of children and adolescents. To determine the influence of social, personal and treatment-related factors on participation, all patients who were actual treated in the international therapy study EuroNet-PHL-C2 in all of Germany (N ≈ 700) and their parents will be interviewed. Statistical analyses will be done using descriptive and multivariate methods taking account of treatment-related issues (e.g. stage of disease, chemotherapy, radiotherapy, progression/relapse).

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed primary diagnosis of classical Hodgkin's Lymphoma
* 10-18 years
* written informed consent of the patient and/or the patient's parents or guardian according to national laws

Exclusion Criteria:

* other (simultaneous) malignancies

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with hodgkin-lymphoma and their parents
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Social participation | one month after diagnosis until two years
  The Child and Adolescent Scale of Participation, CASP
Quality of life | one month after diagnosis until two years
  Questionnaire to assess Health Related Quality of Life in chronically ill Children and Adolescents, KINDL

SECONDARY OUTCOMES:
Understanding of illness | one month after diagnosis until two years
  Illness Perception Questionnaire, IPQ
Autonomy | one month after diagnosis until two years
  Subscale Autonomy from the Health-Related Quality of Life Questionnaire for Children and Adolescents, Kidscreen
Self-efficacy | one month after diagnosis until two years
  Self-Efficacy for Managing Chronic Disease 6-Item Scale, SES6
Optimism | one month after diagnosis until two years
  Subscale from The Bern Subjective Well-Being Questionnaire for Adolescents, BFW
Coping | one month after diagnosis until two years
  Coping Questionnaire for Children and Adolescents, CODI
Sense of coherence | one month after diagnosis until two years
  Children Sense of Coherence Scale, C-SOC
Behavioural disorders and strengths | one month after diagnosis until two years
  Strengths and Difficulties Questionnaire, SDQ
Fatigue | one month after diagnosis until two years
  Subscale Fatigue from the Questionnaire to assess Quality of Life of Cancer Patients developed by the European Organisation for Research and Treatment of Cancer, EORTC QLQ-C30
Satisfaction with treatment | one month after diagnosis until two years
  Questionnaire to assess the Satisfaction with the Treatment, FBB
Social support | one month after diagnosis until two years
  Social Support Scale, SSS

OTHER OUTCOMES:
Parental coping with chronic childhood disease | one month after diagnosis until two years
  Coping Health Inventory for Parents, CHIP (parental questionnaire)
Consequences of chronic conditions and disability in childhood and adolescence for the family | one month after diagnosis until two years
  Impact on Family Scale in Families with Children with Disabilities, FaBel (parental questionnaire)
Family atmosphere | one month after diagnosis until two years
  Family Environment Scale, FES (parental questionnaire)
Psychosocial needs | one month after diagnosis until two years
  Short-Form Supportive Care Needs Survey Questionnaire, SCNS-SF34 (parental questionnaire)
Use of psychosocial care services | one month after diagnosis until two years
  (parental questionnaire)
Satisfaction with treatment | one month after diagnosis until two years
  Questionnaire to assess the Satisfaction with the Treatment, FBB (parental questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Richter, Prof. PhD, Study Chair — Institute of Medical Sociology, Martin Luther University Halle-Wittenberg; Dieter Körholz, Prof. MD, Study Chair — Center for Pediatrics and Adolescent Medicine, Justus-Liebig University of Giessen